CLINICAL TRIAL: NCT05155761
Title: Identifying Risk Factors for Falls in Patients With a High Risk of Fracture Using Connected Insoles (FeetMe Monitor® Device)
Acronym: FAIR
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: FeetMe (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: FTM_FAIR
Record Dates: First submitted 2021-09-15; First posted 2021-12-14 (Actual); Last update posted 2023-06-07 (Actual); Status verified 2023-06

CONDITIONS: Fall; Fall Patients; Osteoporosis
Keywords: FeetMe; Insoles; Fall; Osteoporosis
MeSH Terms: conditions — Osteoporosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Osteoporotic patients (Experimental)
  Interventions: Device: FeetMe® Monitor

INTERVENTIONS:
Device: FeetMe® Monitor — Each patient will be asked to go to 3 visits at the Cochin hospital, and to wear the soles after each of these visits during 3 days, at home, to record the data, so that it reflects walking patterns of the patient in his/her daily life and activities.
  At each visit, clinical tests to assess fall risk will be performed (Timed Up and Go test, one foot stance, Short Physical Performance Battery and 6 minutes walking test ).
  The patients will be supplied with a pair of FeetMe® Monitor insoles, return home and walking parameters will be recorded for 3 to 10 consecutive days.

SUMMARY:
The objective of this study is to determine which gait parameters measured at home using e FeetMe® Insoles are associated with a risk for falls in a patient population suffering from osteoporosis and a higher with high risk of fractures and falls.

Each patient will be asked to go to 3 visits at the Cochin hospital, and to wear the soles after each of these visits during 3 days, at home, to record the data, so that it reflects walking patterns of the patient in his/her daily life and activities.

At the eachvisit, clinical tests to assess fall risk will be performed (Timed Up and Go test, one foot stance, Short Physical Performance Battery and 6 minutes walking test ).

The patients will be supplied with a pair of FeetMe® Monitor Insoles, return home and walking parameters will be recorded for 3 to 10 consecutive days.

ELIGIBILITY:
Inclusion Criteria:

* male and female subjects aged 60 years and above
* with a high fracture and fall risk defined by osteoporosis (low-trauma fracture within the last 5 years and/or osteoporotic bone density)
* a fall within the last year, who own a smartphone.

Exclusion Criteria:

* cognitive deficit or concomitant disorder limiting communication or participation in the study
* simultaneous participation in another study
* deprivation of liberty due to a legal or administrative decision
* patients receiving psychiatric care
* adults beyond the age of majority under legal protection measures or unable to express their consent
* patients admitted to a health or social establishment for reasons other than research.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2021-03-25 (Actual); Primary Completion 2024-11-25 (Estimated); Study Completion 2024-11-25 (Estimated)

PRIMARY OUTCOMES:
To assess how a walking speed decrease at baseline during a 6MWT as measured by the connected Insoles, connected insoles devices, has an effect on risk of fall in subjects with osteoporosis. | at baseline
  Assess walking speed decrease during 6MWT at baseline

CONTACTS AND LOCATIONS:
Locations (1):
- Service de Rhumatologie, Hôpital Cochin, Assistance Publique - Hôpitaux de, Paris, France